CLINICAL TRIAL: NCT03127943
Title: Pilot Study: Comparison of Buffered 1% vs. Non-Buffered 1% Lidocaine Used in Dental and Oral Surgical Procedures: Clinical Outcomes Mandible
Brief Title: Clinical Outcomes Mandible: Buffered 1% vs. Non-Buffered 1% Lidocaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0068
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2018-04

CONDITIONS: Anesthesia, Local
Keywords: lidocaine, mandible
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buffered 1% lidocaine (Active Comparator): In week One, Each subject would be injected intraorally with either anesthetic (Buffered 1% lidocaine with 1/100,00 epinephrine) or (Non-buffered 1% lidocaine with 1/100,00 epinephrine to block the Inferior alveolar, Lingual and Buccal nerves.
  At least a week later injections for the same nerves would involve the alternate anesthetic. Mandibular molar and canine tested for pulpal anesthesia.
  Interventions: Drug: Lidocaine
- Non-buffered 1% lidocaine (Active Comparator): In week Two, Each subject would be injected intraorally with the alternate anesthetic (Buffered 1% lidocaine with 1/100,00 epinephrine) or (Non-buffered 1% lidocaine with 1/100,00 epinephrine to block the Inferior alveolar, Lingual and Buccal nerves.
  At least a week later injections for the same nerves would involve the alternate anesthetic. Mandibular molar and canine tested for pulpal anesthesia.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Efficacy for mandibular molar and canine anesthesia
  Other Names: xylocaine

SUMMARY:
Assess the clinical impact of Buffered 1% lidocaine with epinephrine as compared to the Non-buffered 1% lidocaine with epinephrine in dental and oral surgical procedures.

DETAILED DESCRIPTION:
Background:

Based on the discovery of its topical and locally injected anesthetic effects at the end of the 19th century, cocaine was rapidly adopted as a means of blocking painful sensory impulses from the periphery during surgical procedures.(1) In the last decade local anesthetics have been administered more often, alone or in combination with IV or inhalation anesthetics for most surgical procedures. For clinical procedures in the head and neck the local anesthetic drugs have been combined with a vasoconstrictor, usually epinephrine, to prolong the anesthetic effect at the locally injected anatomic site. To achieve pulpal and periosteal anesthesia by nerve or field block for procedures in dentistry, lidocaine at a 2% concentration has been preferred by clinicians for its reliable outcomes. To prolong the shelf life of the vasopressor, the drug combination must be formulated with a low pH, approximately pH 3.5 for lidocaine with 1/100k epinephrine (Epi).

With a better understanding of the pharmacology, new options for improving local anesthetic effectiveness including buffering the commercially supplied drugs to a neutral pH just prior to injection, continue to emerge.(2) When injected, the low pH causes the "sting" felt by patients on injection. Buffering to a neutral pH eliminates this discomfort and makes the maximum concentration of the non-ionized form of the anesthetic drug immediately available to the targeted nerve membrane.(3-7) Until recently, buffering local anesthetics containing Epi followed with bicarbonate just prior to injection was impractical for the quantities used in intraoral procedures. However, today we do have options to efficiently accomplish this buffering technique.(Anutra Medical, Research TrianglePark, NC).

Buffering local anesthetics just prior to use produces positive outcomes including less "sting" on injection, faster onset of the drug, and possibly added drug potency, ie the same positive clinical effect at lower dosage. In pilot studies with healthy adults as their own controls investigators have shown that Buffered 1% lidocaine with 1/100k Epi was as effective as Non-buffered 2% lidocaine with 1/100k Epi for pulpal anesthesia on a 1st molar or canine after nerve block in the mandible or field block in the maxilla-Phase one of this study.(8,9) These outcomes could be beneficial for performing multiple procedures in children whose lidocaine dosage is limited by body weight or others with chronic liver disease.

Rationale:

The recently reported results from the two clinical studies involving buffered lidocaine with Epi have led to clinicians questioning whether the Buffered 1% lidocaine with Epi might be as effective for achieving pulpal and periosteal anesthesia for dental procedures as Non-Buffered 1% lidocaine with Epi-Phase two of this study, outcomes not usually considered by most clinicians. This protocol addresses that question.

Specific Aims:

Compare clinical depths of pulpal anesthesia for maxillary(Phase one) and mandibular(Phase two) molar and canine teeth at 30min intervals Post-injection of lidocaine Assess pain levels during injection Assess time after injection to lower lip numb

Hypotheses:

No differences exist in anesthetic depth for pulpal anesthesia after intraoral injection mandibular nerve block between Buffered 1% lidocaine with 1/100k epinephrine as compared to Non-buffered 1% lidocaine with 1/100k epinephrine.

Subjects will serve as their own controls in a cross-over AB/BA study design which is uniform within sequences, uniform within periods, and balanced

ELIGIBILITY:
Inclusion Criteria:

Age 18-30 years American Society Anesthesiologists I,II

Exclusion Criteria:

Allergy to lidocaine class of anesthetic drugs Local anesthetic drug use in past week Current symptoms in teeth or oral mucosa

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Turvey, DDS, Study Chair — UNC Oral and Maxillofacial Surgery; Raymond P White Jr, DDS, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Buffered 1% Lidocaine, Then Non-Buffered 1% Lidocaine; Non-Buffered 1% Lidocaine, Then Buffered 1% Lidocaine: At each treatment visit participants were injected to block the Inferior alveolar, Lingual and Buccal nerves.
Period: First Intervention
Arm/Group | Buffered 1% Lidocaine, Then Non-Buffered 1% Lidocaine | Non-Buffered 1% Lidocaine, Then Buffered 1% Lidocaine
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Buffered 1% Lidocaine, Then Non-Buffered 1% Lidocaine | Non-Buffered 1% Lidocaine, Then Buffered 1% Lidocaine
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Buffered 1% Lidocaine, Then Non-Buffered 1% Lidocaine | Non-Buffered 1% Lidocaine, Then Buffered 1% Lidocaine
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were to receive either Buffered 1% lidocaine or Non-Buffered 2% Lidocaine
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [22.5 to 25.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Pulpal Response After Mandibular Molar Anesthesia
Description: Subjects' mandibular molar teeth will be tested before anesthetic and every 30 minutes with cold and electric pulp test for presence of anesthesia as reported by subjects yes or no
Time Frame: Every 30 minutes up to 120 minutes Total
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Buffered 1% Lidocaine, Then Non-Buffered 1% Lidocaine: All subjects who received Buffered 1% Lidocaine
- Non-buffered 1% Lididocaine, the Buffered 1% Lidocaine: All subjects who received Non_buffered Lidocaine
Arm/Group | Buffered 1% Lidocaine, Then Non-Buffered 1% Lidocaine | Non-buffered 1% Lididocaine, the Buffered 1% Lidocaine
Number analyzed (Participants) | 24 | 24
minutes | 100 (37.2) | 106 (41.5)

2. Primary Outcome: Mean Time to Pulpal Response After Mandibular Canine Anesthesia
Description: as for outcome 1
Time Frame: 30 minute intervals up to 120 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Buffered 1% Lidocaine, Then Non-Buffered 1% Lidocaine | Non-buffered 1% Lididocaine, the Buffered 1% Lidocaine
Number analyzed (Participants) | 24 | 24
minutes | 81.3 (44.7) | 97.5 (43.6)

ADVERSE EVENTS:
Time Frame: Every 30 minutes up to 120 minutes total
Groups:
- Buffered 1% Lidocaine: Each subject was injected intraorally with Buffered 1% Lidocaine (with 1/100,00 epinephrine) to block the Inferior alveolar, Lingual, and Buccal nerves. Mandibular molar and canine tested for pulpal anesthesia.
- Non-Buffered 1% Lidocaine: Each subject was injected intraorally with Non-buffered 1% Lidocaine (with 1/100,00 epinephrine) to block the Inferior alveolar, Lingual and Buccal nerves. Mandibular molar and canine tested for pulpal anesthesia.
Arm/Group | Buffered 1% Lidocaine | Non-Buffered 1% Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT03127943/Prot_SAP_000.pdf